CLINICAL TRIAL: NCT00446940
Title: Dose Finding Trial of Rosuvastatin and Atorvastatin Versus Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bader, Ted, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13133
Record Dates: First submitted 2007-03-11; First posted 2007-03-13 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosuvastatin
Drug: atorvastatin

SUMMARY:
Different Doses of rosuvastatin and atorvastatin will be used to see if HCV viral load changes and liver tests change.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C

Exclusion Criteria:

* HIV positivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-12; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Bader, MD, Principal Investigator — VA Medical Center, Oklahoma City, OK
Locations (1):
- VA Hospital, Oklahoma City, Oklahoma, United States